CLINICAL TRIAL: NCT03210688
Title: Treatment of Primary Minimal Change Nephropathy: A Randomized Open-labeled Non-inferiority Study on Prednisolone and Vitamin D
Brief Title: Active Vitamin D And Reduced Dose Prednisolone for Treatment in Minimal Change Nephropathy
Acronym: ADAPTinMCN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADAPT in MCN
Record Dates: First submitted 2017-07-03; First posted 2017-07-07 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Minimal Change Disease; Nephrotic Syndrome
Keywords: Prednisolone; alfacalcidol; Minimal change nephropathy
MeSH Terms: conditions — Nephrosis, Lipoid; Nephrotic Syndrome | interventions — Prednisolone; Prednisone; alfacalcidol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose prednisolone (Active Comparator): Prednisolone 1 mg/kg/day
  Interventions: Drug: Prednisolone
- Alfacalcidol and low dose prednisolone (Experimental): Alfacalcidol 0,5 microgram/day and Prednisolone 0,5 mg/kg/day
  Interventions: Drug: Prednisolone; Drug: Alfacalcidol

INTERVENTIONS:
Drug: Prednisolone — Tablet prednisolone
  Other Names: Prednisone
Drug: Alfacalcidol — Capsule alfacalcidol 0,5 microgram/day
  Arms: Alfacalcidol and low dose prednisolone

SUMMARY:
Traditionally MCN is treated with a high dose of prednisolone, which induces remission in 60-90% of patients. Prednisolone treatment contains numerous side effects and the current dose is empiric. Given the lack of efficacy evidence and the risk associated with the currently accepted treatment regimen there is a need to characterize the outcome in MCN further, and to establish new, and potentially less toxic treatment regimens.

The aim is to examine if treatment with reduced dose of prednisolone in combination with activated vitamin D is as effective as standard high dose prednisolone in achieving remission and preventing relapse in MCN, and if reduced dose prednisolone is associated with fewer side effects compared to standard dose. Furthermore, the study will examine the influence of prednisolone metabolism on the efficacy and side effects of prednisolone in the treatment of MCN.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven minimal change nephropathy
* If earlier minimal change: No relapse in 5 years, and earlier only treated with prednisolone
* Nephrotic syndrome
* Age more than 18 years

Exclusion Criteria:

* Cancer except from basal cells carcinoma
* Lymphoproliferative disease
* Pregnancy
* eGFR < 30 ml/min/1,73m2 (CKD-EPI)
* Allergy
* No danish language
* No ability to give informed prove

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Remission | 4 to 16 weeks
  Time from treatment to remission and the frequency of patients reaching remission on treatment

SECONDARY OUTCOMES:
Relapse | 4 weeks to 1 year after remission
  Frequency of relapse
Side effects to treatment | 4 weeks to 1 year after remission
  The side effects to prednisolone are assessed using questionnaires by both patients and doctors, including SF36 and Cushing QoL. The Glucocorticoid Toxicity Index will be used to quantitate prednisolone-related morbidity.
Concentration of Prednisolone in saliva | 4 weeks after initiating prednisolone treatment
  Measurement of prednisolone metabolism by saliva test and genetic analysis of specific liver enzymes
Rates of genetic polymorphism, including HLA variations | Blood test at baseline
  Genomic HLA typing (HLA-class I: A, B and C and HLA-class II: DM, DO, DP, DQ and DR) will be performed to examine if specific HLA-alleles are more frequent in patients with MCN. Potential modifying genes that theoretically have pathophysiological impact on MCN will be sequenced using targeted next generation sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Per Ivarsen, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Azukaitis K, Palmer SC, Strippoli GF, Hodson EM. Interventions for minimal change disease in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2022 Mar 1;3(3):CD001537. doi: 10.1002/14651858.CD001537.pub5. PMID 35230699
- [Derived] Kristensen T, Birn H, Ivarsen P. A randomised controlled unblinded multicentre non-inferiority trial with activated vitamin D and prednisolone treatment in patients with minimal change nephropathy (ADAPTinMCN). Trials. 2021 Jul 12;22(1):442. doi: 10.1186/s13063-021-05393-4. PMID 34247632